CLINICAL TRIAL: NCT00520221
Title: Intrapleural Minocycline Following Simple Aspiration for Initial Treatment of Primary Spontaneous Pneumothorax: a Retrospective Study
Brief Title: Intrapleural Minocycline Following Simple Aspiration for Primary Spontaneous Pneumothorax
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Other Study IDs: 200707015R
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2004-01

CONDITIONS: Pneumothorax
Keywords: minocycline; pleurodesis; aspiration; pneumothorax; Primary spontaneous pneumothorax; First attack; Successful aspiration
MeSH Terms: conditions — Pneumothorax; cyclopia sequence

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2: Minocycline group: 300 mg of minocycline hydrochloride was instilled into the pleural space through the catheter.
  Control group consisted of 33 patients who had successful simple aspiration alone between January 2004 and December 2005.

SUMMARY:
The optimal initial management of primary spontaneous pneumothorax (PSP) remains controversial. This study was conducted to evaluate the safety and efficacy of additional minocycline pleurodesis after successful aspiration of the first episode of PSP.

DETAILED DESCRIPTION:
Primary spontaneous pneumothorax (PSP) most commonly occurs in young, tall, lean males. The estimated recurrence rate is 23-50% after the first episode. The high recurrence rate stimulated the development of many different therapeutic approaches, ranging from conservative treatment such as observation to more invasive therapies such as surgery, and optimal treatment of patients presenting with a first episode of PSP remains controversial. In the recently published British Thoracic Society (BTS) guidelines, simple aspiration is recommended as the first line treatment for all PSP requiring intervention because this treatment provided the advantage of reduced hospital admission rate and reduced length of hospital stay when compared with chest tube drainage. However, the recurrence rate of this procedure was around 30%, making it inappropriate as a standard of care.

Intrapleural instillation of a chemical irritant (chemical pleurodesis) is an effective way to reduce the rates of recurrent spontaneous pneumothorax in surgical and non-surgical patients. Previously, chemical pleurodesis had usually been administrated through chest tube or thoracoscopy. Administration of sclerosing agents through intravenous needle catheter or pigtail catheter after simple aspiration had never been reported and the safety and efficacy remained unknown.

Because the recurrence rate after simple aspiration remains high, we began to instill minocycline into the pleural cavity through the pigtail or intravenous needle catheter since December 2005 to determine if this adjuvant is effective in reducing the rate of recurrence. In the present study, we report our experience of minocycline pleurodesis in treating first episode of PSP after successful aspiration of pneumothorax. The effects of this adjuvant therapy were evaluated by comparing the outcomes of the patients who underwent simple aspiration alone with those who underwent additional minocycline pleurodesis.

ELIGIBILITY:
Inclusion Criteria:

* Primary spontaneous pneumothorax patients who underwent manual aspiration as their initial treatment were selected.

Exclusion Criteria:

* Patients with a previous history of spontaneous pneumothorax, >50 years of age, or with preexisting pulmonary diseases were excluded. Patients with unsuccessful aspiration requiring further chest tube insertion or thoracoscopic operation were also excluded

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2004-01; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Chie Lee, MD, PhD, Study Chair — Department of Surgery, National Taiwan University Hospital, Taiwan; Jin-Shing Chen, MD, PhD, Study Director — Department of Surgery, National Taiwan University Hospital, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan